CLINICAL TRIAL: NCT05879965
Title: Prospective On-site and Questionnaire Study for the FOLLOW-UP of Mpox Cohort at ITM PLUS Evaluation of the Longevity of B- and T-cell Immune Responses in Former Mpox Patients and Vaccine Recipients
Brief Title: Prospective Study for the FOLLOW-UP of Human Monkeypox Cases and Smallpox Vaccinees at Risk
Acronym: POQS-FU PLUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 1628/22
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Monkeypox
Keywords: mpox; immunology; mucosal immunity; sequelae; smallpox vaccination
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, PBMC, saliva, semen, anal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mpox patients: mpox cohort diagnosed and confirmed by PCR at the Institute of Tropical Medicine (ITM) in Antwerp during the recent mpox outbreak May-October 2022, 95 consented patients for follow-up
- Smallpox vaccine recipients: sub-group 1: 100 participants routinely vaccinated with two subcutaneous 3rd generation smallpox vaccines sub-group 2: 100 participants routinely vaccinated with two intradermal 3rd generation smallpox vaccines
- Healthy controls: 50 controls recruited during HIV-PrEP consultation (no former mpox infection, no smallpox vaccination)

SUMMARY:
The goal of this observational study is to describe possible physical and psychological sequelae after an mpox infection and to evaluate the longevity of B- and T-cell immune responses in former mpox patients and vaccine recipients.

The main questions it aims to answer are:

* Are there any physical or pschological sequelae after mpox infection?
* Is the humoral and/or cellular immune response to MPOX (or vaccinia) virus) durable?
* Do the patients develop strong local immunity in comparison to systemic immunity?
* How long is the virus still detectable in semen, saliva or the ano-rectal region?

Participants will answer a questionnaire, samples with blood, saliva and semen as well as anal swabs will be collected. Follow-up visits 8, 16 and 24 months after infection or vaccination are planned.

A healthy control group will be recruited in our HIV-PrEP clinic.

DETAILED DESCRIPTION:
Long-term problems or sequelae after an acute viral infection are described. The study aim is to investigate if long-term symptoms and sequelae can be found in the ITM human mpox infection cohort previously diagnosed and confirmed by PCR at the Institute of Tropical Medicine in Antwerp during the mpox outbreak 2022 in Belgium. The immune response after a natural mpox infection and after a smallpox vaccination will additionally analysed over time.

Consented participants Mpox patients, acute infection (n=169, 21% assumed smallpox vaccination in childhood) Mpox patients for follow-up (n=95, 20% assumed smallpox vaccination in childhood) Smallpox vaccinees, two intradermal doses (n=100) Smallpox vaccinees, two subcutaneous doses (n=100) Healthy unvaccinated controls (n=50)

Design This prospective longitudinal study has the main objectives to describe possible physical and psychological sequelae after an mpox infection and to evaluate the longevity of B- and T-cell immune responses in former mpox patients and vaccine recipients. Participants are being followed up 8, 16 and 24 months after infection or vaccination.

Sample collection Anal eSwabs from patients, controls and vaccinees Saliva (Omnigene-oral and dry swabs) from patients, controls and vaccinees Serum from patients, controls and vaccinees Optional semen samples from patients PBMC samples from a sub-group of patients, controls and vaccinees

Laboratory analysis MPXV-PCR on saliva, anorectal and optional semen samples of former mpox patients, vaccinated individuals and healthy controls Mpox-specific antibody profiling from serum Mucosal immunity (IgA, IgG) mpox-specific/reactive from anal swabs and/or saliva Enumeration of MPXV-specific effector-memory T cells via flow cytometry-based AIM or ICS assays (peptide pool stimulation or HLA-restricted multimer-based capture assays) Enumeration of MPXV-specific memory B cells or plasma cells via flow cytometry-ased AIM or ICS assays (recombinant antigen stimulation or HLA-restricted multimer-based capture assays)

ELIGIBILITY:
Mpox patients for immunological study

Inclusion criteria

* PCR-confirmed monkeypox infection since May 2022
* ≥18 years
* Willingness to provide written informed consent
* Willingness to follow the study schedule

Exclusion criteria

* Born before 1976
* Any documented or remembered smallpox vaccination or typical scar for a smallpox vaccination
* Any vaccination 2 weeks before or after the visits (4 weeks for life-vaccines)
* Any immune-compromising drugs or diseases (treated and controlled HIV-infection is no exclusion criteria)
* Any mpox reinfection since study start

Smallpox vaccinees for immunological study

Inclusion criteria

* Two 3rd generation smallpox vaccinations either two subcutaneous or two intradermal vaccinations with a minimum of 4 weeks and a maximum of 8 weeks interval. First vaccination given after 01 August 2022.
* ≥18 years
* Willingness to provide written informed consent
* Willingness to follow the study schedule

Exclusion criteria

* Born before 1976
* Any documented or remembered smallpox vaccination or typical scar for a smallpox vaccination
* Any vaccination 2 weeks before or after the visits (4 weeks for life-vaccines)
* Any immune-compromising drugs or diseases (treated and controlled HIV-infection is no exclusion criteria)
* Any mpox infection in the past

HIV-Prep patients

Inclusion criteria

* On HIV-PrEP and a patient from ITM
* ≥18 years
* Willingness to provide written informed consent
* Willingness to follow the study schedule

Exclusion criteria

* Born before 1976
* Any documented or remembered smallpox vaccination or typical scar for a smallpox vaccination
* Any vaccination 2 weeks before or after the visits (4 weeks for life-vaccines)
* Any immune-compromising drugs or diseases
* Any mpox infection in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former mpox patients ≥18 years, diagnosed by PCR at ITM since May 2022 Smallpox vaccine recipients (2xSC) or (2xID), routinely vaccinated at ITM since August 2022 Healthy HIV-PrEP users
Sampling Method: Non-Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with a positive mpox serology in both groups | 2 years
  To compare the MPXV-specific serological response in naturally infected mpox male patients 8, 16 and 24 months after onset of symptoms with the MPXV-specific serological response in routinely (=2 either subcutaneous (SC) or intradermal (ID) vaccinations with an interval of 4-8 weeks) vaccinated men against smallpox 8 months after the first vaccination
Proportion of long-term problems or sequelae in mpox patients | 2 years
  To describe any possible long-term problem or sequela after an acute human mpox infection diagnosed and confirmed by PCR at ITM since the beginning of the mpox outbreak End of May 2022

SECONDARY OUTCOMES:
longevity of humoral and/or cellular immune response to mpox or vaccinia virus | 2 years
  B-cell and T-cell characteristics in former mpox patients and smallpox vaccinees 8, 16, 24 months after symptom

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Berens-Riha, PhD, Principal Investigator — Institute of Tropical Medicine; Laurens Liesenborghs, PhD, Study Director — Institute of Tropical Medicine
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided